CLINICAL TRIAL: NCT06553300
Title: Auto Transplantation of Wisdom Teeth With or Without Platelet Rich Fibrin for Replacement of Non-Restorable Posterior Teeth.
Brief Title: Auto Transplantation of Wisdom Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDIOS00011
Record Dates: First submitted 2024-07-29; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Autotransplantation of Wisdom Teeth; Patelet Rich Fibrin
MeSH Terms: interventions — Transplantation, Autologous; Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autotransplantation with PRF (Experimental)
  Interventions: Procedure: Autotransplantation with PRF
- Autotrasplantation only (Active Comparator)
  Interventions: Procedure: Autotransplatation Only

INTERVENTIONS:
Procedure: Autotransplantation with PRF — Autotransplantation of Wisdom teeth to the extracted socket of removed broken down posterior teeth with the application of PRF
  Arms: Autotransplantation with PRF
Procedure: Autotransplatation Only — Autotransplantation of Wisdom teeth to the extracted socket of removed broken down posterior teeth.
  Arms: Autotrasplantation only

SUMMARY:
Autotransplantation emerges as a viable alternative to tooth extraction and prosthetic restoration when conventional endodontic treatments are unfeasible or contraindicated. The success of autotransplantation is influenced by diverse factors, including root development stage, tooth morphology, surgical technique, extraoral duration, recipient socket shape, recipient bed vascularity, and periodontal ligament cell vitality. Preserving periodontal ligament quality and achieving tissue adaptation are pivotal for successful tooth transplantation. Successful donor tooth replacement is influenced by variables like fitting attempts, alveolus-root distance, extra-alveolar time, surgical skill, and extraction trauma intensity.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* aged between 20 and 50 years
* devoid of systemic ailments
* complying with the study procedures
* holding an Anesthesiologists classification of 1 or 2
* possessing mandibular or maxillary immature wisdom teeth

Exclusion Criteria:

* systemic diseases that might impede the healing process
* Patients with pacemakers
* Individuals harboring allergies to medications or antibiotics
* active smokers
* patients afflicted with periodontal diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic success | one year
  The success of auto-transplanted immature third molars with and without Platelet-Rich Fibrin will be assessed over a year period.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Elmallah, DDS, Study Chair — Cleveland Dental; Ahmed Hashem, DDS, Study Director — Cleveland Dental
Locations (1):
- Cleveland Dental Institute, Cleveland, Ohio, United States